CLINICAL TRIAL: NCT01128075
Title: Multi-center, Two-arm Non-comparative, Observational, 96-week Phase IV Study to Evaluate Treatment Adherence When Using RebiSmart™ for Self-injection of Rebif® in Multi-dose Cartridges in Subjects With Relapsing Multiple Sclerosis (RMS)
Brief Title: Treatment Adherence When Using RebiSmart™ in Relapsing Multiple Sclerosis Subjects
Acronym: MEASURE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: EMD Inc., Canada (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR701068-520
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis; MS
Keywords: RebiSmart; Rebif; Adherence; Multidose; Relapsing Multiple Sclerosis; RMS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- naïve subjects: Cohort of RMS patients who initiate disease modifying treatment with Rebif®
  Interventions: Device: RebiSmart™
- non-naïve subjects: Cohort of RMS patients who initiate treatment with Rebif® after having failed therapy with other disease modifying drugs on the basis of lack of efficacy, compliance, safety, tolerability or convenience, as per clinical judgment of study investigator
  Interventions: Device: RebiSmart™

INTERVENTIONS:
Device: RebiSmart™ — Electronic self-injection device (RebiSmart™) to inject Rebif®
  Other Names: Rebif
  Groups: naïve subjects
Device: RebiSmart™ — Electronic self-injection device (RebiSmart™) to inject Rebif®
  Other Names: Rebif
  Groups: non-naïve subjects

SUMMARY:
This is a multi-center, two-arm non-comparative, observational, 96 week Phase IV study to evaluate treatment adherence when using RebiSmart™ for self-injection of Rebif® in subjects with relapsing multiple sclerosis (RMS).

Subjects who have a confirmed diagnosis of RMS using McDonald Criteria and meet the eligibility criteria during a screening period of up to 28 days will be provided with an electronic self-injection device (RebiSmart™) to inject Rebif® for 96 weeks.

The main purpose of this study is to evaluate treatment adherence for subjects with RMS over 24 weeks of treatment when using RebiSmart™ for self-injection of Rebif® in a multi-dose cartridge.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age.
* Have RMS according to the revised McDonald Criteria.
* Subject is eligible for Rebif® therapy according to indications and clinical use in the Rebif® Product Monograph.
* Be willing and able to comply with the protocol requirements for the duration of the study.
* Have given written informed consent prior to entering the screening period.
* Must register with the Rebif® Multiple Support Program.
* Subjects previously on disease modifying drugs (DMDs) must be stable and not be experiencing any side effects related to the previous DMDs at the time of enrollment into the study, in the opinion of the investigator. Rebif® will be prescribed as per Product Monograph and a washout period will be left at the discretion of the investigator.

Exclusion Criteria:

* Have any disease other than MS that could better explain his/her signs and symptoms.
* Receive any other injectable medications on a regular basis during the week prior to the screening period or throughout the duration of the study. The administration of a single injection for treatment or prophylaxis of a condition unrelated to the subject's MS (e.g.,influenza or pneumococcus vaccination) will be acceptable.
* Are contraindicated for the use of Rebif® according to the Rebif® Product Monograph.
* Have a diagnosis of clinically isolated syndrome (CIS).
* Participation in any other investigational trial prior to 30 days of Study Day 1.
* Any visual or physical impairment that precludes the subject from self-injecting the treatment using RebiSmart™
* Have received previous treatment with Rebif within 5 years prior to screening.
* Subjects have any medical, psychiatric or other conditions that compromise his/her ability to understand the subject information, to give informed consent, to comply with the study protocol or to complete the study questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community and Academic MS clinics
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2009-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Treatment adherence for RMS subjects over 24 weeks of treatment when using RebiSmart™ for self-injection of Rebif® in a multi-dose cartridge. | 24 weeks

SECONDARY OUTCOMES:
Long-term adherence in subjects with RMS over 96 weeks of treatment using RebiSmart for self-injection of Rebif® in multi-dose cartridge. | 96 weeks
Treatment persistence by measuring treatment discontinuations | 96 weeks
Treatment compliance | 96 weeks
  Measuring the number of injections received relative to the time on study
Comparison of subject treatment adherence between categories of cognitive function | 96 weeks
  Measured by the short version of Rao's Brief Repeatable Battery (BRB)
Longitudinal changes in anxiety symptoms | 96 weeks
  Measured by the Hospital Anxiety and Depression Scale (HAD) and State-Trait Anxiety Inventory (STAI)
Qualitative assessment of subjects' experience with RebiSmart | 96 weeks
  A standardized Patient Experience Questionnaire (PEQ) will be used for the assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, a division of EMD Inc., Canada
Locations (1):
- University of British Columbia, Vancouver, Canada

REFERENCES:
- [Derived] Devonshire VA, Feinstein A, Moriarty P. Adherence to interferon beta-1a therapy using an electronic self-injector in multiple sclerosis: a multicentre, single-arm, observational, phase IV study. BMC Res Notes. 2016 Mar 8;9:148. doi: 10.1186/s13104-016-1948-z. PMID 26951043